CLINICAL TRIAL: NCT04789850
Title: Safety and Efficacy of Itacitinib in Adults With Systemic Sclerosis: a Phase II, Randomized, Controlled Trial
Brief Title: Safety and Efficacy of Itacitinib in Adults With Systemic Sclerosis
Acronym: SCLERITA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP180613; 2019-003430-16 (EudraCT Number)
Record Dates: First submitted 2021-02-10; First posted 2021-03-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Itacitinib
MeSH Terms: conditions — Scleroderma, Systemic | interventions — itacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itacitinib (Experimental): 200mg of oral Itacitinib everyday for 360 days.
  Interventions: Drug: Itacitinib
- Placebo (Placebo Comparator): Oral placebo everyday for 360 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itacitinib — 200 mg oral for 360 days
  Arms: Itacitinib
Drug: Placebo — 200 mg oral for 360 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether itacitinib is safe and effective in the treatment of systemic sclerosis in adults.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare systemic autoimmune connective tissue-disease characterized by fibrosis, inflammation, and vasculopathy. SSc is responsible for skin fibrosis that can either be limited or diffuse. The latter phenotype of the disease is commonly associated with visceral involvement and therefore similar to graft versus host disease (GvHD) reaction. It can be life threatening in case of pulmonary or cardiovascular involvement. Nonetheless SSc remains a severe disease responsible for important disability and a poor quality of life.

There is a growing body of evidence that supports the implication of the JAK-STAT tyrosine kinases pathway in the activation of fibroblasts of patients with SSc. A genetic polymorphism of STAT4 was found to be associated with the diffuse form of the disease and inhibition of STAT4 gene is associated with a decrease in TGF-ß and IL-6 cytokines activation, which are two major cytokines implicated in SSc pathogenesis. Recently, Pedroza et al. confirmed the implication of STAT3 in skin fibrosis mechanisms. Indeed, the authors showed an enhanced activation of STAT3 and demonstrated in vivo that the inhibition of STAT3 phosphorylation prevented skin fibrosis in a murine model of SSc. These data were confirmed by a work of Zhang et al. who showed that the inhibition of JAK1 was also needed to prevent skin and lung fibrosis. Altogether these works confirmed the implication of the JAK pathway in fibrosis mechanism.

Itacitinib is a Janus kinase inhibitor that specifically targets JAK1 and decreases STAT3 phosphorylation. Itacitinib was shown to efficiently treat patients with myelofibrosis, rheumatoid arthritis, and chronic plaque psoriasis. Very interestingly, itacitinib efficacy has also been reported in patients with acute GvHD. Altogether these data and studies reinforced the investigator's working hypothesis.

The efficacy and safety of this proposal must be tested.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Patient with a diagnosis of diffuse SSc, as defined by the American College of Rheumatology / EULAR 2013 criteria,
* Patient with a diffuse SSc, according to Leroy and Medsger dichotomy
* Patient with a SSc disease duration of less than 36 months (defined as time from first non-Raynaud phenomenon manifestation) or with an active SSc disease, as defined by EUSTAR disease activity score,
* Patient with a modified Rodnan skin score (mRSS) ≥ 10 and ≤ 35 units at screening,
* Negative pregnancy test for woman of childbearing potential, woman of childbearing potential should have reliable contraception for the 12 months' duration of the study,
* Patient able to give written informed consent prior to participation in the study,
* Affiliation to a social security scheme (profit or being entitled)
* If patients receive mycophenolate or methotrexate for SSc, these need to be on stable dose as follows:

  * Mycophenolate mofetil/sodium: stable dose for at least 2 months prior to randomisation
  * Methotrexate: stable dose and route of administration for at least 2 months prior to randomisation

Exclusion Criteria:

* Previous treatment with itacitinib or a Janus kinase (JAK) inhibitor,
* Contra-indications to itacitinib or Janus kinase inhibitor,
* Failure to sign the informed consent or unable to consent
* Patient participating in another investigational therapeutic study,
* Acute or chronic active infections, including HBV, HCV, HIV,
* Patient with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patient suspected not to be observant to the proposed treatments,
* Patient who have white blood cell count ≤ 4,000/mm3,
* Patient who have platelet count ≤ 100,000/mm3,
* Patients who have ALT or AST level greater that 3 times the upper limit of normal,
* Patient who have triglyceride level greater than 5g/L
* Pregnant or breastfeeding woman,
* Protected adults (including individual under guardianship by court order),
* Patient receiving or having received cyclophosphamide or rituximab within the last three months (possible inclusion beyond 3 months),
* Patient receiving or having received a biotherapy (anti-TNF, abatacept or tocilizumab) in the last 3 months (possible inclusion beyond 3 months)
* Patient with Systemic Lupus, or Sjögren's syndrome with systemic manifestations justifying immunosuppressive therapy
* Atherosclerotic cardiovascular disease as defined by a history of myocardial infarction, ischaemic stroke, or peripheral artery thrombosis
* Anti-phospholipid syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) at 360 days | 360 days
  performed by the same investigator at day 0 and day 360 and the change in mRSS will be calculated following the formula: ΔmRSS= mRSSd360 - mRSSd0.
  To measure mRSS, skin thickness of the patient is rated by palpation at each of 17 anatomic sites using a scale of 0-3 (0 = normal skin; 1= mild thickness; 2= moderate thickness; 3=severe thickness with an inability to pinch the skin into a fold). The scores at each site are summed with a minimum of 0 and a maximum of 51 (17 sites)

SECONDARY OUTCOMES:
Incidence of death | at 180 and 360 days
Incidence of Adverse Events | at 180 and 360 days
  according to the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading scale
Incidence of Severe Adverse Events | at 180 and 360 days
  according to the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading scale
Change in modified Rodnan skin score at 90, 180, 270 days | at 90, 180 and 270 days
Proportion of patients who improved mRSS at 90, 180, 270 and 360 days | At 90, 180, 270 and 360 days
Proportion of patients with an active disease according to the European scleroderma trials and research group (EUSTAR)SSc activity score at 90, 180, 270 and 360 days | At 90, 180, 270 and 360 days
  EUSTAR SSc activity index score from 0 to 10 - a cut-off ≥ 2.5 identifies patients with active disease
Change in the Combined Response Index in Diffuse Systemic Sclerosis (CRISS) score | At 180 and 360 days
  composite response index
SSc disease activity | At 90, 180, 270 and 360 days
  * Physicians visual analogue scale range from 0 (min) to 10 (max) - 0=no activity, 10=maximum activity
  * Patients visual analogue scale range from 0 (min) to 10 (max) - 0=no activity, 10=maximum activity
Short Form-36 (SF-36) health questionnaire | At 0, 15, 90, 180, 270 and 360 days
  self-administered questionnaire of 36 items assessing the following 8 domains : physical functioning, bodily pain, role limitations attributable to physical health problems, general health perceptions, mental health, role limitations to emotional problems, vitality and social functioning (scale from 0 to 100)
EurolQol-5Domain (EQ-5D) health questionnaire | At 0, 15, 90, 180, 270 and 360 days
  self reported measure of quality of life - (scale from 0 to 100)
Health Assessment Questionnaire Disability Index (HAQ-DI) scale | At 0, 15, 90, 180, 270 and 360 days
  self administered 20 questions- score range from 0 (no disability) to 3 (severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Mouthon, MD-PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Benjamin Chaigne, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (42):
- France (42):
  - CH Amiens, Amiens
  - CHU Angers, Angers
  - CHU Annecy, Annecy
  - CHU Besançon, Besançon
  - Avicenne Hospital, Bobigny
  - CHU Bordeaux, Bordeaux
  - Ambroise Paré hospital, Boulogne-Billancourt
  - Hôpital de la Cavale Blanche, Brest
  - CHU Caen, Caen
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Henry Mondor hospital, Créteil
  - CH Dax-Côte d'ARgent, Dax
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon sud, Lyon
  - Hôpital Nord, Marseille
  - La Timone Hospital, Marseille
  - Robert Schuman Hospital, Metz
  - CHU Montpellier - rhumatology, Montpellier
  - CHU Montpellier - St Eloi Hospital, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hopital L'Archet 1, Nice
  - Hospital Pasteur - CHU Nice, Nice
  - Saint Antoine Hospital, Paris
  - La Pitié-Salpêtrière, Paris
  - Cochin Hospital, Paris
  - Hospital Croix St Simon, Paris
  - CHU Poitiers, Poitiers
  - CH de Cornouaille, Quimper
  - Robert Debré Hospital, Reims
  - Hôpital Sud, Rennes
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Nouvel Hospital Civil, Strasbourg
  - Rangueil Hospital, Toulouse
  - CHU Tours, Tours
  - CH Valenciennes, Valenciennes
  - Hôpitaux de Barbois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Almeida C, Almeida I, Vasconcelos C. Quality of life in systemic sclerosis. Autoimmun Rev. 2015 Dec;14(12):1087-96. doi: 10.1016/j.autrev.2015.07.012. Epub 2015 Jul 23. PMID 26212726
- [Background] Mouthon L. SSc in 2011: From mechanisms to medicines. Nat Rev Rheumatol. 2012 Jan 10;8(2):72-4. doi: 10.1038/nrrheum.2011.203. PMID 22231235
- [Background] Distler JH, Feghali-Bostwick C, Soare A, Asano Y, Distler O, Abraham DJ. Review: Frontiers of Antifibrotic Therapy in Systemic Sclerosis. Arthritis Rheumatol. 2017 Feb;69(2):257-267. doi: 10.1002/art.39865. No abstract available. PMID 27636741
- [Background] Wang Y, Fan PS, Kahaleh B. Association between enhanced type I collagen expression and epigenetic repression of the FLI1 gene in scleroderma fibroblasts. Arthritis Rheum. 2006 Jul;54(7):2271-9. doi: 10.1002/art.21948. PMID 16802366
- [Background] Landi C, Bargagli E, Bianchi L, Gagliardi A, Carleo A, Bennett D, Perari MG, Armini A, Prasse A, Rottoli P, Bini L. Towards a functional proteomics approach to the comprehension of idiopathic pulmonary fibrosis, sarcoidosis, systemic sclerosis and pulmonary Langerhans cell histiocytosis. J Proteomics. 2013 May 27;83:60-75. doi: 10.1016/j.jprot.2013.03.006. Epub 2013 Mar 23. PMID 23528693
- [Background] Kubo M, Ihn H, Yamane K, Tamaki K. Up-regulated expression of transforming growth factor beta receptors in dermal fibroblasts in skin sections from patients with localized scleroderma. Arthritis Rheum. 2001 Mar;44(3):731-4. doi: 10.1002/1529-0131(200103)44:33.0.CO;2-U. No abstract available. PMID 11263790
- [Background] Zhang Y, Liang R, Chen CW, Mallano T, Dees C, Distler A, Reich A, Bergmann C, Ramming A, Gelse K, Mielenz D, Distler O, Schett G, Distler JHW. JAK1-dependent transphosphorylation of JAK2 limits the antifibrotic effects of selective JAK2 inhibitors on long-term treatment. Ann Rheum Dis. 2017 Aug;76(8):1467-1475. doi: 10.1136/annrheumdis-2016-210911. Epub 2017 May 6. PMID 28478401
- [Background] Migita K, Izumi Y, Torigoshi T, Satomura K, Izumi M, Nishino Y, Jiuchi Y, Nakamura M, Kozuru H, Nonaka F, Eguchi K, Kawakami A, Motokawa S. Inhibition of Janus kinase/signal transducer and activator of transcription (JAK/STAT) signalling pathway in rheumatoid synovial fibroblasts using small molecule compounds. Clin Exp Immunol. 2013 Dec;174(3):356-63. doi: 10.1111/cei.12190. PMID 23968543
- [Background] Xu Y, Wang W, Tian Y, Liu J, Yang R. Polymorphisms in STAT4 and IRF5 increase the risk of systemic sclerosis: a meta-analysis. Int J Dermatol. 2016 Apr;55(4):408-16. doi: 10.1111/ijd.12839. Epub 2015 Dec 29. PMID 26712637
- [Background] Avouac J, Furnrohr BG, Tomcik M, Palumbo K, Zerr P, Horn A, Dees C, Akhmetshina A, Beyer C, Distler O, Schett G, Allanore Y, Distler JH. Inactivation of the transcription factor STAT-4 prevents inflammation-driven fibrosis in animal models of systemic sclerosis. Arthritis Rheum. 2011 Mar;63(3):800-9. doi: 10.1002/art.30171. PMID 21360510
- [Background] Kremer JM, Bloom BJ, Breedveld FC, Coombs JH, Fletcher MP, Gruben D, Krishnaswami S, Burgos-Vargas R, Wilkinson B, Zerbini CA, Zwillich SH. The safety and efficacy of a JAK inhibitor in patients with active rheumatoid arthritis: Results of a double-blind, placebo-controlled phase IIa trial of three dosage levels of CP-690,550 versus placebo. Arthritis Rheum. 2009 Jul;60(7):1895-905. doi: 10.1002/art.24567. PMID 19565475
- [Background] Fridman JS, Scherle PA, Collins R, Burn T, Neilan CL, Hertel D, Contel N, Haley P, Thomas B, Shi J, Collier P, Rodgers JD, Shepard S, Metcalf B, Hollis G, Newton RC, Yeleswaram S, Friedman SM, Vaddi K. Preclinical evaluation of local JAK1 and JAK2 inhibition in cutaneous inflammation. J Invest Dermatol. 2011 Sep;131(9):1838-44. doi: 10.1038/jid.2011.140. Epub 2011 Jun 16. PMID 21677670
- [Background] Deverapalli SC, Rosmarin D. The use of JAK inhibitors in the treatment of progressive systemic sclerosis. J Eur Acad Dermatol Venereol. 2018 Aug;32(8):e328. doi: 10.1111/jdv.14876. Epub 2018 Mar 6. No abstract available. PMID 29444362
- [Background] Gordon JK, Martyanov V, Franks JM, Bernstein EJ, Szymonifka J, Magro C, Wildman HF, Wood TA, Whitfield ML, Spiera RF. Belimumab for the Treatment of Early Diffuse Systemic Sclerosis: Results of a Randomized, Double-Blind, Placebo-Controlled, Pilot Trial. Arthritis Rheumatol. 2018 Feb;70(2):308-316. doi: 10.1002/art.40358. Epub 2017 Dec 29. PMID 29073351